CLINICAL TRIAL: NCT07164625
Title: The Effectiveness of Telerehabilitation vs. In-person Physiotherapy in Young Elite Baseball Players With Rotator Cuff Pathology: A Randomized Controlled Trial
Brief Title: Telerehabilitation vs. In-person Physiotherapy in Young Elite Baseball Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE22241A
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Tendinopathy
Keywords: rotator cuff tear; rotator cuff tendinopathy; telerehabilitation; baseball
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): A 6-week program delivered via real-time video sessions
  Interventions: Behavioral: Telerehabilitation Physiotherapy
- In-person (Active Comparator): A 6-week program delivered face-to-face, including hands-on treatments
  Interventions: Behavioral: In person physiotherapy

INTERVENTIONS:
Behavioral: Telerehabilitation Physiotherapy — Delivered via real-time video sessions focusing on strengthening and mobility exercises.
  Arms: Telerehabilitation
Behavioral: In person physiotherapy — face-to-face, including hands-on treatments like tactile feedback and joint mobilization.
  Arms: In-person

SUMMARY:
This study compares physical therapy delivered through video calls to in-person therapy for young baseball players with shoulder pain. The goal is to see if remote therapy is as effective and easier for them to stick with

DETAILED DESCRIPTION:
This study compares physical therapy delivered through video calls to in-person therapy for young baseball players with shoulder pain. The goal is to see if remote therapy is as effective and easier for them to stick with

ELIGIBILITY:
Inclusion Criteria:

* unilateral shoulder symptoms (chronic pain, instability, or weakness) for more than 3 months together with a diagnosis of rotator cuff tendinopathy or mild partial-thickness tear (≤25% of tendon thickness) confirmed by ultrasound or MRI

Exclusion Criteria:

* history of prior shoulder surgery within the past 12 months; partial-thickness tear greater than 25% or full-thickness tear; associated pathology requiring surgical management (e.g., humeral head avulsion fracture); significant elbow symptoms or injury; systemic inflammatory disease; neurologic disorders affecting upper limb function; and inability to comply with the intervention or scheduled assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Kerlan-Jobe Orthopaedic Clinic (KJOC) Shoulder and Elbow Score | 6 weeks
  Change in scores on the KJOC, a self-reported questionnaire assessing functional performance in overhead athletes.

SECONDARY OUTCOMES:
Pain Intensity | 6 weeks
  Measured by a Visual Analogue Scale (VAS) on a scale from 0 (no pain) to 10 (most painful)
Shoulder painless range of motion (ROM) | 6 weeks
  Abduction, external rotation, and internal rotation
Isokinetic External Rotation (ER) Strength | 6 weeks
  Measured at 60°/s and 180°/s with Biodex

OTHER OUTCOMES:
Supervised Session Attendance | 6 weeks
  Percentage of attended sessions out of 12 at 6 weeks.
Home Exercise Compliance | 6 weeks
  Percentage of completed sessions based on self-reported logs at 6 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taichung, Taiwan